CLINICAL TRIAL: NCT02519712
Title: Treatment of Elderly AML Patients With Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells From Haploidentical Related Donors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-141
Record Dates: First submitted 2015-08-06; First posted 2015-08-11 (Estimated); Results first posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2017-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Induction Chemotherapy; G-CSF-Mobilized Stem Cells; Haploidentical Related Donors; 15-141
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Induction Chemotherapy

ARMS (1):
- Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells (Experimental): This is a single center trial to assess the feasibility of standard induction chemotherapy followed by a single dose of unmanipulated G-PBSC for the treatment of elderly patients with newly diagnosed AML.
  Interventions: Drug: Induction Chemotherapy; Procedure: G-PBSC Infusion

INTERVENTIONS:
Drug: Induction Chemotherapy — Patients with newly diagnosed AML will receive standard induction chemotherapy with daunorubicin and cytarabine (7+3 scheme). Patients who achieve CR may undergo consolidation chemotherapy at the discretion of the treating leukemia physician.
Procedure: G-PBSC Infusion — G-CSF-mobilized peripheral blood cells will be collected from the donors in the Donor Room according to standard MSKCC BMT guidelines. Patients will be infused by infusion of unmanipulated G-PBSC from a haploidentical related donor.

SUMMARY:
The purpose of this study is to test a method of bone marrow transplantation that results in only temporary donor immune function. In other words, the donor immune cells are given in a way that will allow them to attack leukemia briefly before being destroyed by their own immune system, or "rejected." The investigators want to test whether temporary donor immune function is enough to improve the odds of achieving a remission without exposing the patient to the toxicities of a full bone marrow transplant. To do this, the investigators will use standard chemotherapy for AML followed by an infusion of donor stem cells. The donor will be a family member who is haploidentically, or half matched, to the patient such as a child or sibling. Chemotherapy designed to treat AML should not be strong enough to prevent them from rejecting the donor stem cells. The investigators will then follow the patient to see how long the donor stem cells stay in them. The study will test whether this process is feasible and can result in improved chances of obtaining a remission.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60.
* Patients with a new diagnosis of histologically confirmed (according to WHO classification 2008) acute myeloid leukemia (either primary or secondary AML) are included.
* Patients with a diagnosis of myelodysplastic syndrome with >/= 10% bone marrow blasts with no response or progression of disease after at least 4 cycles of a hypomethylating agent (5-azacytiine or decitabine).
* Patients must have a healthy blood-related donor (parent, child, sibling) willing to undergo apheresis after G-CSF administration.
* Karnofsky performance status > 70%.
* Hepatic function - total bilirubin < 2 and, AST < 2.5 x upper limit of normal, unless liver is involved with disease or a history of Gilbert's disease.
* Renal function - adequate renal function as demonstrated by a serum creatinine <2 mg/dl.
* LVEF ≥ 50% as determined by echocardiogram or MUGA.
* Ability to give informed consent.

Donor Eligibility:

* Donor is blood-related and HLA-haploidentical to the recipient.
* Donor ≥18 years old
* Donor has undergone serologic testing for transmissible diseases as per blood banking guidelines for organ and tissue donors. Tests include but are not limited to: HepBsAg, HepBsAb, HepBcAb, HepC antibody, HIV, HTLV I and II, VZV, CMV and VDRL, and West Nile Virus . Donor must have normal negative test results for HIV, HTLV I and II, and West Nile Virus.
* Donor has a CXR and EKG performed.
* Donor is not allergic to G-CSF.
* Donor must be able to undergo leukapheresis
* Donor is not pregnant.
* Donor does not have concurrent malignancy or autoimmune disease.
* Ability to give informed consent.

Exclusion Criteria:

* Patients with a diagnosis of acute promyelocytic leukemia (according to WHO classification 20080
* Major surgery or irradiation within two weeks.
* Previous therapy with cytotoxic agents for AML. Persons with previous treatments for myelodysplasia/myeloproliferation such as hydroxyurea, interferon, hypomethylating agents (5-azacitidine or decitabine), lenalidomide, or JAK/STAT inhibitors may participate but must have >1 week off therapy prior to enrollment.
* Active CNS disease.
* Uncontrolled infection.
* Pregnant or lactating women - they are excluded, given the potential teratogenic effects of chemotherapy and agents used in the therapy.
* Male and female patients of child-bearing potential unwilling to use effective means of contraception.
* HIV or HTLV I/II seropositivity.
* Concurrent active malignancy other than AML requiring therapy.
* Clinically significant cardiac disease (NY Heart Association Class III or IV) or pulmonary disease.
* Inability or unwillingness to comply with the treatment protocol, follow-up, or research tests

Donor Exclusion:

* Donor has cardiac risk factors precluding ability to undergo leukapheresis.
* Donor has evidence of concurrent malignancy or autoimmune disease.
* Donor is pregnant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shaffer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells: This is a single center trial to assess the feasibility of standard induction chemotherapy followed by a single dose of unmanipulated G-PBSC for the treatment of elderly patients with newly diagnosed AML.
  Donors and participants are combined because the study was closed to poor accrual and there are no clinical results.
Period: Overall Study
Arm/Group | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells
Started | 4
Completed | 0
Not Completed | 4
Not completed — Disease Relapse | 1
Not completed — Disease Progression | 1
Not completed — Accruals are donors | 2

BASELINE CHARACTERISTICS:
Groups:
- Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells: This is a single center trial to assess the feasibility of standard induction chemotherapy followed by a single dose of unmanipulated G-PBSC for the treatment of elderly patients with newly diagnosed AML.
  Adverse Events information cannot be separated by donors and recipients due to data privacy reasons.
Arm/Group | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: Peripheral Blood Counts: The peripheral blood neutrophil count should be ≥1,500/μl (sustained without growth factor support), and the platelets count should be ≥100,000/μl (without transfusion). No circulating blasts (in the absence of growth factor) should be detected.
  Bone Marrow Aspirate: The cellularity of the bone marrow should approximate normal. There must be evidence of maturation of all cell lines. The bone marrow aspirate should contain < 5% blasts. Auer rods should not be detected.
  Extramedullary Leukemia: Extramedullary leukemia, such as CNS or soft tissue involvement, must not be present.
Time Frame: 4 weeks
Population: Data were not collected
Arm/Group | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Discharge to 100 +/- 7 days
Arm/Group | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells
All-Cause Mortality (participants affected / at risk) | 2/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells (N=4)
Abdominal Pain (Gastrointestinal disorders) | 2
Platelet count decreased (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Chemotherapy Followed by G-CSF-Mobilized Stem Cells (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02519712/Prot_SAP_000.pdf